CLINICAL TRIAL: NCT02326519
Title: Electrical Signal Collection From a 20 Pole Catheter During Routine Cardiac Procedures
Acronym: E20PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E20PC study
Record Dates: First submitted 2014-12-10; First posted 2014-12-29 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intracardiac electrode catheter (Other): All patient in the study will have same data collected during the procedure using the Steerable intracardiac electrode catheter.
  Interventions: Other: Intracardiac electrode catheter

INTERVENTIONS:
Other: Intracardiac electrode catheter — All patient in the study will have the same data collected using the Steerable intracardiac electrode catheter

SUMMARY:
Routine data collection will be conducted during normal sinus rhythm and AV synchronous pacing for approximately 20 minutes. The data collected will then be processed and the P, R and T wave amplitudes will be measured.

DETAILED DESCRIPTION:
The purpose of this study is to collect atrio-ventricular electrograms using a sequence of tip-ring spacings in patients undergoing routine cardiac procedures (EP study, pacemaker/ICD/CRT implant). To collect these signals, a 20 pole catheter (Medtronic StableMapr intracardiac steerable electrode catheter) will be acutely placed in the RV apex during a routine cardiac procedure.

Routine data collection will be conducted during normal sinus rhythm and AV synchronous pacing for approximately 20 minutes. The data collected will then be processed and the P, R and T wave amplitudes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or above, or of legal age to give consent specific to the national law of the countries in which the study is being conducted

  * Subjects who are undergoing a cardiac procedure where routine placement of cardiac catheter can be performed
  * Subjects are willing to provide Informed Consent

Exclusion Criteria:

* • Subject has exclusion criteria per local law and regulations (e.g. age, breast feeding, etc)

  * Any condition which precludes the subject's ability to comply with the study requirements
  * Subject has physical conditions that contraindicate the use of the device per approved labeling, including but not limited to active sepsis, known sensitivity to heparin, cannot undergo standard anticoagulation protocol for cardiac procedure, blood clotting abnormalities or a recent coagulopathy or embolic event, venous filtering device (Greenfield Filter) and obstructed or damaged vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-01-13 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
The electrical signal mean amplitude (mv) during AV synchronous pacing. | 2 minutes during the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Allgemeines Krankenhaus der Stadt Linz, Linz, Austria
- Hôpital Cardiologique du Haut-Lévêque, Bordeaux, France